CLINICAL TRIAL: NCT00674232
Title: Misoprostol for Treatment of Incomplete Abortion
Brief Title: Treatment of Incomplete Abortion With 600 Mcg Oral Misoprostol Compared to Standard Surgical Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Dr. Beverly Winikoff, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.2.0
Record Dates: First submitted 2008-04-28; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Incomplete Abortion
Keywords: incomplete abortion; spontaneous miscarriage
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol; Surgical Procedures, Operative; Dilatation and Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Experimental): Group 1 randomized to take single dose of 600 mcg oral misoprostol
  Interventions: Drug: 600 mcg misoprostol
- Surgical treatment (Other): Group 2 randomized to receive standard surgical treatment as per local protocol (D&C or MVA)
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Drug: 600 mcg misoprostol — single dose of misoprostol taken orally
  Other Names: Cytotec
  Arms: Misoprostol
Procedure: Surgical treatment — Either dilation and curettage or manual vacuum aspiration, as per local protocol
  Other Names: D&C, MVA
  Arms: Surgical treatment

SUMMARY:
This study aims to compare the efficacy, side effects profile and acceptability of a single dose of 600mcg misoprostol taken orally compared to standard surgical treatment as per local protocols for the treatment of incomplete abortion.

ELIGIBILITY:
Inclusion Criteria:

* past or present history of vaginal bleeding during pregnancy
* open cervical os
* evidence of incomplete abortion with substantial debris in the uterus (if using ultrasound)
* surgical evacuation of the uterus would be advised as course of action if misoprostol was not available
* generally in good health
* woman lives or works within one hour of study site
* woman willing to provide contact information for follow up purposes
* informed consent given

Exclusion Criteria:

* contraindications to study drug
* uterine size larger than 12 weeks LMP
* signs of severe infection

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2006-05; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
complete resolution of signs/symptoms of incomplete abortion without recourse to surgery at any point for any reason | one week after initial treatment

SECONDARY OUTCOMES:
side effects | measured at follow up visit one week after initial treatment
acceptability | measured at follow up visit one week after initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Peña, MPH, MA, Study Director — Gynuity Health Projects; Jill Durocher, Study Director — Gynuity Health Projects
Locations (3):
- Ecuador (2):
  - Hospital del Dia, CEMOPLAF, Quito
  - Hospital Gineco-obstetrico Isidro Ayora, Quito
- Hospital Maternidad Concepcion Palacios, Caracas, Venezuela

REFERENCES:
- [Derived] Montesinos R, Durocher J, Leon W, Arellano M, Pena M, Pinto E, Winikoff B. Oral misoprostol for the management of incomplete abortion in Ecuador. Int J Gynaecol Obstet. 2011 Nov;115(2):135-9. doi: 10.1016/j.ijgo.2011.06.015. Epub 2011 Aug 26. PMID 21872244
- See also: Related Info — http://www.gynuity.org